CLINICAL TRIAL: NCT03145454
Title: Objective Markers of Pain Perception in Pediatric Emergency
Acronym: TAMALOU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1608198; ANSM (Other: 2017-A00340-53)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Suffering, Physical
Keywords: Pain; children; emergency; electroencephalography; heart rate; skin conductance; pupillary diameter
MeSH Terms: conditions — Pain; Emergencies | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain detection (Experimental): Electroencephalographical responses will be collected during surgical gesture by different intervention: electroencephalography helmet, dermal electrode, blood pressure sensors, pupillometry glasses and Holter.
  Interventions: Device: electroencephalography helmet; Device: dermal electrode; Device: blood pressure sensors; Device: Pupillometry glasses; Device: Holter

INTERVENTIONS:
Device: electroencephalography helmet — electroencephalography helmet with twelve electrodes will be performed during surgical gesture to determine the pain of child.
Device: dermal electrode — dermal electrode on the back of the hand will be performed during surgical gesture to determine the pain of child.
Device: blood pressure sensors — blood pressure sensors on the finger will be performed during surgical gesture to determine the pain of child.
Device: Pupillometry glasses — Pupillometry glasses will be performed during surgical gesture to determine the pain of child.
Device: Holter — Three electrodes electrocardiography on the chest will be performed during surgical gesture to determine the heart rate variability.

SUMMARY:
Pain is a major problem in the care of children in pediatric emergencies. Indeed, its relief rests on the oral communication of the young patient, who does not always able to it (difficult to verbalize, fear of the hospital, problem mental development ...). There is no way in which pain can be apprehended objectively, immediately and effectively. To advance our knowledge of this problem, several approaches have been studied as from functional magnetic resonance imaging (fMRI), electroencephalography (EEG), or from autonomic parameters. However, all these approaches have their limitations: although fMRI presents interesting performances, it allows only a retrospective analysis, and cannot adapt to the clinical context of the young patient for example. EEG-based approaches and autonomic parameters show interesting results but suffer from perfectible sensitivity to muscle activation for EEG whereas the vegetative parameters to stress. In this context, our working hypothesis considers that the search for markers of painful perception must be based on a neurophysiological approach, based on the combined analysis of the EEG and autonomic responses in real time. The aim of this work is to study (1) the cortical (EEG) and autonomic (cardiovascular, skin, pupillary) responses induced by sutures in children who can communicate their pain according to whether they cause pain or not.

ELIGIBILITY:
Inclusion Criteria:

* Requiring one or more non-complex sutures in department of pediatric emergency
* Affiliate or beneficiary of social security (parents)
* Signature of consent (parents)

Exclusion Criteria:

* Historic of cardiovascular diseases (arterial hypertension, etc), renal or metabolic syndrome (diabetes etc.), psychiatric (depression, etc.) or neurological (epilepsy seizure, etc.)
* Trouble of heart rhythm
* Allergy at conductive gel for electrode
* Sutures requiring a general anesthesia
* Contraindication at the Xylocaine and/or Paracetamol

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Measure of alpha spectral power | During the surgical gesture
  Compare measures of alpha spectra power according to electroencephalography helmet and electrode electrocardiography results.

SECONDARY OUTCOMES:
Rate of spectral power low and high frequency | During the surgical gesture
  Rate of spectral power low and high frequency according to heart frequency variability result.
Amplitude of the dermal responsiveness | During the surgical gesture
  Compare amplitude of the dermal responsiveness according to dermal electrode result.
Amplitude of the pupillary diameter | During the surgical gesture
  Compare amplitude of the pupillary diameter according to pupillometry glasses result.

CONTACTS AND LOCATIONS:
Overall Officials: Hugues PATURAL, MD PhD, Principal Investigator — CHU SAINT-ETIENNE; Florian CHOUCHOU, PhD, Study Chair — SAINT-ETIENNE UNIVERSITY
Locations (1):
- Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No